CLINICAL TRIAL: NCT00308295
Title: A Pilot Study of Fish Oil Supplementation in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0512-13
Record Dates: First submitted 2006-03-27; First posted 2006-03-29 (Estimated); Last update posted 2007-10-16 (Estimated); Status verified 2007-10

CONDITIONS: End-Stage Renal Disease Patients on Hemodialysis
MeSH Terms: interventions — Fish Oils

INTERVENTIONS:
Drug: Fish oil capsules
Drug: matched placebo capsules

SUMMARY:
The main goal of this study is to determine whether the American Heart Association-recommended fish oil dose is efficacious, safe, and tolerable in hemodialysis patients. The secondary objective is to test the effects of fish oil supplementation on inflammatory and cardiovascular markers.

ELIGIBILITY:
Exclusion Criteria:

1. Age <18
2. Pregnant individuals
3. Fish oil or omega-3 supplementation in past 6 months
4. Fish, corn, soybean, gelatin, or vanilla allergies
5. Currently enrolled in a dietary or investigational drug study
6. Life expectancy < 3 months
7. Ongoing active illness requiring hospitalization
8. Malabsorption syndromes
9. Chronic heparin or coumadin anticoagulation (??)
10. Active bleeding issues

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27
Dates: Start 2006-04; Study Completion 2006-05

PRIMARY OUTCOMES:
To determine whether AHA-recommended fish oil therapy beneficially affects the pro-inflammatory/anti-inflammatory blood fatty acid balance

SECONDARY OUTCOMES:
To test the safety and tolerability of fish oil therapy in hemodialysis patients
To measure the effects of fish oil treatment on cardiovascular and inflammatory risk factors

CONTACTS AND LOCATIONS:
Overall Officials: Allon Friedman, MD, Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - Indiana University Nephrology Clinics, Indianapolis, Indiana
  - VeteransAdministration Hospital, Indianapolis, Indiana